CLINICAL TRIAL: NCT01152476
Title: Emergency Agitation in T&A
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: professor, Seoul National University Bundang Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: T&A_EA
Record Dates: First submitted 2010-06-25; First posted 2010-06-29 (Estimated); Last update posted 2011-01-06 (Estimated); Status verified 2011-01

CONDITIONS: Healthy
Keywords: healthy pediatric patients undergoing tonsillectomy and adenoidectomy
MeSH Terms: interventions — Remifentanil; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- group SR (Active Comparator)
  Interventions: Drug: remifentanil
- group S (Active Comparator)
  Interventions: Drug: normal saline

INTERVENTIONS:
Drug: remifentanil — General anesthesia is maintained witn sevoflurane and remifentanil.
  Arms: group SR
Drug: normal saline — General anesthesia is maintained with only sevoflurane and with normal saline instead of remifentanil
  Arms: group S

SUMMARY:
Sevoflurane has been used commonly in pediatric anesthesia since 1990. However, it has caused more emergency agitation (EA) that other inhalation agents and the incidence is up to 80%. Therefore, lower minimum alveolar concentration of sevoflurane will reduce the EA when it is used with remifentanil in pediatric general anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologist physical status I or II
* 2-6 year-old children
* patients undergoing tonsillectomy and adenoidectomy

Exclusion Criteria:

* upper respiratory disease
* mental retardation

Ages: 2 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 42 (Estimated)
Dates: Start 2010-04; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
emergency agitation | during 1 hour after recovering of anesthesia
  at post-anesthetic care unit

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea